CLINICAL TRIAL: NCT02502240
Title: Frequency of ALK Rearrangements in Non Small-Cell Lung Cancer in Latin America: The Latin-American Consortium for the Investigation of Lung Cancer (CLICaP).
Brief Title: ALK Rearrangements in Lung Adenocarcinoma: Epidemiology in Latin America (CLICaP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, Master of biological sciences, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: ALK-CLICaP
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Lung Cancer
Keywords: ALK; Latin American
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of the frequency and clinical characteristics of ALK rearrangements in Latin-American countries.

Latin American countries are heterogeneous in terms of lung cancer incidence, ethnicity, and exposure to potential carcinogens. The discovery of the echinoderm microtubule-associated protein like 4-anaplastic lymphoma kinase (EML4-ALK) translocation as an oncogenic driver has led to the development of novel therapies with activity in vitro and in the clinic.

DETAILED DESCRIPTION:
The precise frequency of ALK in Latin American population has not been determined. Studies isolated in some Latin American countries like Brazil report a frequency of 3.2%, Argentina of 4.2% and Mexico of 9.0% of ALK fusion in a small number with lung cancer. Reliable information about ALK frequencies and disparities among ethnic groups is critical. Our study pretends to know the frequency and clinical characteristics of ALK rearrangement of Latin American patients with NSCLC. Discusses the difficulty of having a single diagnostic test for this chromosome abnormality.

The development of efficient and reliable laboratory test is critical in the selection of patients likely to respond to these targeted agents. Currently, the current gold standard for testing for EML4-ALK translocation is fluorescent in situ hybridization (FISH) for selecting patients for ALK-tyrosine kinase inhibitors (TKI) therapy according to the United States Food and Drug Administration (FDA). But, an important aspect is the amount of available tumor present in a determined sample, given the labor-intensive nature and cost of the test, there has been interest in validating other screening and diagnostic tools. Recent evidence suggests that ALK Immunohistochemistry (IHC) instruments globally protocols, can be very effective in the detection of ALK rearrangement in NSCLC (ALK+) tumors expressing the fusion ALK protein.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed lung cancer and tissue availability for ALK analysis.

Exclusion Criteria:

* Not lung cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both: both female and male participants are being studied Analysis of the ALK translocation was done either by FISH, IHC, or both, with an adequate amount of cancer cells. Demographic, clinical and pathological data was obtained from patients.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Anaplastic Lymphoma Kinase (ALK) tumor rearrangement status in Non-Small Cell Lung Cancer (NSCLC) patients | 1 year
  Positive or negative status. Evaluated by three diagnostic methods: (1) fluorescence in situ hybridization (FISH), (2) immunohistochemistry (IHC) and (3) real-time polymerase chain reaction (RT-qPCR).

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Gerardo Arrieta Rodriguez, MD MSc, Principal Investigator — Instituto Nacional de Cancerología Mexico city
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takeuchi K, Choi YL, Soda M, Inamura K, Togashi Y, Hatano S, Enomoto M, Takada S, Yamashita Y, Satoh Y, Okumura S, Nakagawa K, Ishikawa Y, Mano H. Multiplex reverse transcription-PCR screening for EML4-ALK fusion transcripts. Clin Cancer Res. 2008 Oct 15;14(20):6618-24. doi: 10.1158/1078-0432.CCR-08-1018. PMID 18927303
- [Background] Lopes LF, Bacchi CE. Anaplastic lymphoma kinase gene rearrangement in non-small-cell lung cancer in a Brazilian population. Clinics (Sao Paulo). 2012 Jul;67(7):845-7. doi: 10.6061/clinics/2012(07)23. No abstract available. PMID 22892933
- [Background] Arrieta O, Cardona AF, Martin C, Mas-Lopez L, Corrales-Rodriguez L, Bramuglia G, Castillo-Fernandez O, Meyerson M, Amieva-Rivera E, Campos-Parra AD, Carranza H, Gomez de la Torre JC, Powazniak Y, Aldaco-Sarvide F, Vargas C, Trigo M, Magallanes-Maciel M, Otero J, Sanchez-Reyes R, Cuello M. Updated Frequency of EGFR and KRAS Mutations in NonSmall-Cell Lung Cancer in Latin America: The Latin-American Consortium for the Investigation of Lung Cancer (CLICaP). J Thorac Oncol. 2015 May;10(5):838-843. doi: 10.1097/JTO.0000000000000481. PMID 25634006